CLINICAL TRIAL: NCT06665347
Title: Effect of Yoga on Psychological Aspect and Quality of Life in Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Arwa Mohamed Abd El-Wahab, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004757
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2024-10

CONDITIONS: Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Autogenic Training; Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive muscle relaxation group (Active Comparator): All participants in this group will receive progressive muscle relaxation for 8 weeks
  Interventions: Other: Progressive muscle relaxation
- Progressive muscle relaxation and Yoga group (Experimental): All participants in this group will receive the same progressive muscle relaxation plus yoga for 8 weeks.
  Interventions: Other: Progressive muscle relaxation; Other: Yoga

INTERVENTIONS:
Other: Progressive muscle relaxation — The participants will receive progressive muscle relaxation for 8 weeks. The muscles of the hand, arm, face, shoulder and neck, chest, abdomen, back, thigh and hip, legs and feet will be contracted and relaxed in sequence. The contraction time is 5 seconds (s), and the relaxation time is 10s.
Other: Yoga — The participants will receive yoga for 30 minutes/session, 3 sessions/week for 8 weeks. The session will begin with 5 minutes for warming up. Twenty minutes of wind relieving position (pavanmuktasana), corpse position (savasana), standing side stretch position, seated forward bend (paschimothanasana), cobra position (bhujangasana), and chair position (utkatasana). Five minutes of cooling down.
  Arms: Progressive muscle relaxation and Yoga group

SUMMARY:
This study will be carried out to evaluate the effect of yoga on psychological aspect and quality of life in premenstrual syndrome.

DETAILED DESCRIPTION:
Premenstrual syndrome (PMS) is characterized by a collection of physical, emotional, psychological, and behavioral symptoms that appear in a cyclic and recurring pattern during the late luteal phase of the menstrual cycle and alleviate within two to four days of menstruation.

Premenstrual Syndrome has a negative impact on young girls' lives, which can lead to reduced work efficiency and quality of work, increased accidents and lack of school attendance. Therefore, there is a need to develop treatment protocols for coping with premenstrual symptoms.

Yoga denotes union and integration and improves biopsychosocial and spiritual wellness. In other words, yoga is a form of mind-body health that combines physical activity with inner-directed mindfulness to achieve self-consciousness through breathing and meditation.

So, this study will be conducted to contribute and add new information that may help the field of physical therapy. It will provide an evidence base for the efficacy of yoga on management of psychological aspect and quality of life in premenstrual syndrome, owing to its low cost, and ease use that may lead to improvement of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Their ages will be ranged from 18 to 25 years old.
* Their body mass index (BMI) will be less than 30 kg/m².
* They will be virgin.
* They will have regular menstrual cycles.
* They will suffer from Premenstrual syndrome based on daily record of severity of problems.
* All women will be conscious and free from any medical disease.

Exclusion Criteria:

* Women with the following criteria should be excluded from this study:
* Women with endocrine disturbance.
* Endometriosis.
* Pelvic inflammatory disease.
* Any pelvic pathology conditions.
* Women had hysterectomy or ovariectomy.
* Women use medications as contraceptive pills, pain relief drugs and antidepressant drugs.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2024-11-02 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of premenstrual symptoms | 8 weeks
  It will be assessed using daily record of severity of problems (DRSP). It was used to capture premenstrual symptoms. DRSP contained two parts: symptoms related to menstruation (21 items) and their impairment in daily life (3 items). The symptoms included depression, hopelessness, feelings of worthlessness, increased sleeping, trouble sleeping, feeling overwhelmed, breast tenderness, breast swelling, headache, joint or muscle pain, anger, conflicts or problems with people, anxiety, mood swings, sensitivity to rejection, decreased interest, difficulty concentrating, fatigue, increased appetite, craving specific foods, and feeling out of control All items were rated from 1 ("not at all") to 6 ("extreme"). The higher the score, the more severe the premenstrual symptoms.
Assessment of anxiety | 8 weeks
  The spielberger state trait anxiety inventory will be used to assess anxiety for all participants. It is a 40-item self-report measure of anxiety using a 4-point Likert-type scale for each item. It has two scales: State anxiety, i.e. how one feels at the moment; and Trait anxiety, i.e. how one generally feels. Both scales consist of 20 items. its score is ranged from 20-80 on both its two subscales.
  from 20-37 means no or low anxiety, 38-44 means moderate anxiety and 45-80 means severe anxiety.
Assessment of depression: | 8 weeks
  It will be assessed using Beck depression inventory. It is a 21-item, self-rated scale that evaluates key symptoms of depression including mood, pessimism, sense of failure, self-dissatisfaction, guilt, punishment, self-dislike, self-accusation, suicidal ideas, crying, irritability, social withdrawal, indecisiveness, body image change, work difficulty, insomnia, fatigability, loss of appetite, weight loss, somatic preoccupation, and loss of libido. its score is ranged from 0-63 and the lowest is zero.
Assessment of Quality of life | 8 weeks
  the SF-36 questionnaire will be used to assess quality of life for all participants. It consists of 36 questions. The SF-36 assesses eight dimensions that include: physical function, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitation due to emotional problems, and mental health. the score is ranged from 0-100. 1 is for the worse health and 100 for the ideal health.
Assessment of stress level | 8 weeks
  A blood sample will be taken from each woman in the two groups at pre-treatment and post-treatment to measure cortisol levels at 8 AM before breakfast for all cases. it will be used as an objective indication of pain level. its normal values are 5 to 25 mcg/dl or 140-690 nmol/L.
Assessment of pain intensity | 8 weeks
  It will be assessed using the visual analogue scale (VAS). VAS is a simple and frequently used method for the assessment of variations in intensity of pain. In clinical practice the percentage of pain relief, assessed by VAS, is often considered as a measure of the efficacy of treatment. the scale ranges from 0 to 10 with 0 meaning no pain and 10 meaning severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Al Din Kamel, Professor, Study Director — Al-Azhar University; khadyga Abdul Aziz, Professor, Study Chair — Cairo University
Locations (1):
- Arwa mohamed Abd El-Wahab, Cairo, Egypt